CLINICAL TRIAL: NCT00975234
Title: Phase II, Randomised, Controlled Study of Treatment With Revascularisation Surgery With or Without Injection of Autologous Skeletal Myoblasts in Patients With Old Myocardial Infarction
Brief Title: Treatment With Autologous Skeletal Myoblasts
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Fina Biotech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mio/Reg/Quirur/Aleatorizado
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Old Myocardial Infarction
Keywords: Intra-lesion injection of autologous myoblasts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skeletal myoblasts (Experimental): Patients who are receiving skeletal myoblasts
  Interventions: Procedure: Intra-lesion injection of autologous skeletal myoblasts; Procedure: Revascularisation
- Placebo (Placebo Comparator): Revascularisation surgery
  Interventions: Procedure: Revascularisation

INTERVENTIONS:
Procedure: Intra-lesion injection of autologous skeletal myoblasts — Intra-lesion injection
  Arms: Skeletal myoblasts
Procedure: Revascularisation — Revascularisation surgery

SUMMARY:
The purpose of this study is to determine the benefit of autologous skeletal myoblast injection in patients with old myocardial infarction and ventricular dysfunction versus conventional revascularisation therapy.

DETAILED DESCRIPTION:
Ischaemic heart disease is one of the main causes of mortality and morbidity. In particular, myocardial infarction (MI) is of special significance, as the heart muscle cannot regenerate so a region's necrosis leads to the formation of a fibrous scar. Depending on the area affected by the scar, infarction can lead to a progressive and irreversible decline in cardiac function, giving way to heart failure (HF) syndrome. The molecular basis of congestive heart failure is the absence of cardiac stem cells capable of regenerating cardiac muscle. In the skeletal muscle, there are cells located beneath the basal membrane with are capable of regenerating muscle fibres; they are known as myoblasts. There are several studies with autologous myoblasts, either by direct administration during surgery or percutaneously, which could distinguish between the effect of revascularisation surgery and that of the myoblast injection. The objective of this study is compare improvement in global and regional cardiac function in patients with old MI obtained by aortocoronary bypass surgery with intracardiac administration of autologous skeletal myoblasts versus standard aortocoronary bypass surgery treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of coronary disease obtained by coronary angiography who require conventional aortocoronary bypass surgery.
* History of myocardial infarction with evidence of regional akinesis (or dyskinesia) for more than 4 weeks and less than 10 years.
* Ejection fraction from 25% to 45%.
* Evidence of no regional viability by dobutamine echocardiography.
* Aged from 30-80 years old.
* Negative serology to HIV, HBV and HCV.
* Patients without organ dysfunction.
* Negative pregnancy test (women of childbearing age).
* Informed consent granted.

Exclusion Criteria:

* History of myocardial infarction in the 4 weeks prior to the inclusion in the study.
* Prior history of tachycardia or ventricular fibrillation (except in patients with DAI device).
* History of cancer (except basocellular carcinoma) or prior treatment with chemotherapy.
* The patient should not suffer from any concomitant severe and/or uncontrolled medical condition.
* Patients who, due to their geographical, psychiatric or social status, have difficulties in meeting the conditions established in the protocol.
* Pregnant or beast feeding women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoints will be evaluate the ejection fraction and wall motion score index measured by M-mode and echocardiography 12 months after surgery. | 12 months after surgery

SECONDARY OUTCOMES:
Secondary efficacy endpoints are viability, perfusion and thickening and incidence of cardiac arrhythmias. | 12 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Prósper, MD, PhD, Study Director — Clinica Universidad de Navarra
Locations (6):
- Spain (6):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital La Fe, Valencia, Valencia